CLINICAL TRIAL: NCT01089569
Title: Evaluation of Insulin Glargine and Exenatide: A Randomized Clinical Trial With Continuous Glucose Monitoring and Ambulatory Glucose Profile Analysis
Brief Title: Continuous Glucose Monitoring Evaluation of Exenatide Twice Daily Versus Insulin Glargine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03951-10-C
Record Dates: First submitted 2010-03-17; First posted 2010-03-18 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; continuous glucose monitoring; exenatide; insulin glargine
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Masking Description: Subjects were randomized and then told the medications they were randomized to. Since the medications were already on the market, there was no need for masking for any involved individuals.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide (Active Comparator): 5 mcg BID (twice daily) for 1 month increasing to 10 mcg BID for the remainder of the study
  Interventions: Drug: Exenatide
- Insulin Glargine (Active Comparator): .1 unit per kg to start, titrated based on Continuous Glucose Monitoring results
  Interventions: Drug: Insulin Glargine
- Exenatide + Insulin Glargine (Active Comparator): Exenatide: 5 mcg BID (twice daily) for 1 month increasing to 10 mcg BID for the remainder of the study
  + Insulin Glargine: 0.1 unit per kg to start, titrated based on Continuous Glucose Monitoring results
  Interventions: Drug: Exenatide; Drug: Insulin Glargine

INTERVENTIONS:
Drug: Exenatide — 5 mcg BID (twice daily) for 1 month increasing to 10 mcg BID for the remainder of the study
  Other Names: Bydureon
  Arms: Exenatide; Exenatide + Insulin Glargine
Drug: Insulin Glargine — .1 unit per kg to start, titrated based on Continuous Glucose Monitoring results
  Other Names: Lantus
  Arms: Exenatide + Insulin Glargine; Insulin Glargine

SUMMARY:
The primary purpose of this study is to compare the effect on 24-hour blood glucose patterns, HbA1c, and weight management when adding insulin glargine, or exenatide, or a combination of insulin glargine and exenatide to metformin.

DETAILED DESCRIPTION:
The primary objective of this study was to characterize the diurnal glucose patterns produced by insulin glargine alone, exenatide (GLP-1 agonist) alone and the combination of insulin glargine and exenatide in subjects taking stable dose of metformin and to evaluate their efficacy in terms of improvement in glucose exposure, variability, stability, incidence of hypoglycemia and weight management.

An ancillary study was approved as part of this study. The purpose of the ancillary study was to use CGM to characterize the glycemic response to a fixed breakfast meal consumed by study participants receiving different medications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥18 and ≤75 years of age
* Clinical diagnosis of type 2 diabetes
* Diabetes duration ≥ 1 year
* HbA1c ≥7.0%
* Currently treated with metformin (HbA1c ≤9%) or metformin/sulfonylurea (SU) (HbA1c ≤8%)or SU alone (HbA1c ≤8%)

Exclusion Criteria:

* Previously treated with insulin or incretin-based therapy
* Treated with a thiazolidinedione within past 6 weeks
* Taken oral or injected prednisone or cortisone medications in the previous 30 days
* Any pancreatic disease or at high risk of pancreatitis (history of alcohol abuse, active gallbladder disease)
* Serum creatinine >1.4mg/dL (women) or >1.5 mg/dL (men)
* eGFR (Estimated Glomerular Filtration Rate) <30 ml/min (using MDRD/ Modification of Diet in Renal Disease equation)
* ALT(Alanine Transaminase) > 2x Upper Limit of Normal (ULN)
* Presence of any severe medical or psychological condition or chronic conditions/infections that in the opinion of the Investigator would compromise he subject's safety or successful participation in the study
* Currently pregnant or planning pregnancy during the study period
* Unable to follow the study protocol
* Unable to speak, read and write in English
* Uncontrolled hyperglycemia with HbA1c > 9% on metformin or >8% on SU or metformin/SU combination or ketonuria requiring immediate insulin therapy
* At the investigator's discretion for other medical or psychological reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet; Roger S Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet; Elinor S Strock, APRN, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mazze RS, Strock E, Wesley D, Borgman S, Morgan B, Bergenstal R, Cuddihy R. Characterizing glucose exposure for individuals with normal glucose tolerance using continuous glucose monitoring and ambulatory glucose profile analysis. Diabetes Technol Ther. 2008 Jun;10(3):149-59. doi: 10.1089/dia.2007.0293. PMID 18473688
- [Background] Mazze R, Strock E, Morgan B, Wesley D, Bergenstal R, Cuddihy R. Diurnal glucose patterns of exenatide once weekly: a 1-year study using continuous glucose monitoring with ambulatory glucose profile analysis. Endocr Pract. 2009 May-Jun;15(4):326-34. doi: 10.4158/EP09046.ORR. PMID 19454385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Started | 20 | 20 | 20
Completed | 16 | 17 | 16
Not Completed | 4 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Exenatide: 5 mcg BID for 1 month increasing to 10 mcg BID for the remainder of the study
  Exenatide: refer to Arm detail
- Insulin Glargine: .1 unit per kg to start, titrated based on Continuous Glucose Monitoring results
  Insulin Glargine: refer to Arm detail
- Total: Total of all reporting groups
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine | Total
Number analyzed (Participants) | 16 | 17 | 16 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.8) | 53.8 (7.4) | 56.7 (8.7) | 56.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 7 | 23
  Male | 10 | 7 | 9 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 17 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change
Description: Measure the changes in HbA1C attributable to exenatide, insulin glargine and their combination.
  Employ CGM with AGP analysis to determine if there is an incremental benefit for subjects who do not reach target to add exenatide to insulin glargine or insulin glargine to exenatide in patients taking metformin.
Time Frame: baseline to final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: %HbA1c
Groups:
- Exenatide: 5 mcg BID for 1 month increasing to 10 mcg BID for the remainder of the study
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
%HbA1c
  Baseline | 6.4 (0.3) | 6.4 (0.5) | 6.2 (0.5)
  Final - Week 32 | 7.8 (.6) | 7.6 (.5) | 7.6 (.7)

2. Secondary Outcome: Change From Baseline in Incidence of Hypoglycemia (Frequency)
Description: Employ Continuous Glucose Monitoring (CGM) with Ambulatory Glucose Profile (AGP) analysis to characterize the diurnal patterns produced by oral medications (metformin) used in the treatment of type 2 diabetes.
  Employ CGM to measure the effect of exenatide, insulin glargine and exenatide plus insulin glargine in terms of underlying physiological defects and alter medications in a manner that improves- iv. Incidence of hypoglycemia (frequency)
  Change from baseline was calculated as mean incidence rate at baseline minus mean incidence rate at final visit (32 weeks)
Time Frame: baseline to final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: episodes/day
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
episodes/day | .7 (0.8) | .8 (0.8) | .6 (0.4)

3. Secondary Outcome: Change From Baseline in Incidence of Hypoglycemia (Degree)
Description: Employ Continuous Glucose Monitoring (CGM) with Ambulatory Glucose Profile (AGP) analysis to characterize the diurnal patterns produced by oral medications (metformin) used in the treatment of type 2 diabetes.
  Employ CGM to measure the effect of exenatide, insulin glargine and exenatide plus insulin glargine in terms of underlying physiological defects and alter medications in a manner that improves- iv. Incidence of hypoglycemia (degree) Change from baseline was calculated as mean incidence percentage at baseline minus mean incidence percentage at final visit (32 weeks)
Time Frame: baseline to final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: percentage of measures under 70 mg/dL
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
percentage of measures under 70 mg/dL | 1.7 (2.7) | 1.7 (1.8) | 1.3 (1.1)

4. Secondary Outcome: Change From Baseline in Glucose Stability (Absolute Hourly Rate of Change in Median Curve)
Description: Employ Continuous Glucose Monitoring (CGM) with Ambulatory Glucose Profile (AGP) analysis to characterize the diurnal patterns produced by oral medications (metformin) used in the treatment of type 2 diabetes.
  Employ CGM to measure the effect of exenatide, insulin glargine and exenatide plus insulin glargine in terms of underlying physiological defects and alter medications in a manner that improves iii. Glucose stability (absolute hourly rate of change in median curve)
  Change from baseline was calculated as mean absolute hourly rate of change in median curve at baseline minus rate at final visit (32 weeks). Mean absolute hourly rate of change in the smoothed median curve is calculated as delta subscript MC = (|p subscript 50 zero - p subscript 50 23|+Sum superscript 23 subscript i = 1| p subscript 50i - p subscript 50 i-1| over T.
  i = hour of day p subscript 50i = smoothed 50th percentile value for ith hour of day T = total # of non-missing hourly smoothed percentiles
Time Frame: baseline to final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL/hr
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
mg/dL/hr | -2 (2.7) | -2.9 (4.4) | -2 (3.5)

5. Secondary Outcome: Change From Baseline in CGM Glucose Variability
Description: Employ Continuous Glucose Monitoring (CGM) with Ambulatory Glucose Profile (AGP) analysis to characterize the diurnal patterns produced by oral medications (metformin) used in the treatment of type 2 diabetes.
  Employ CGM to measure the effect of exenatide, insulin glargine and exenatide plus insulin glargine in terms of underlying physiological defects and alter medications in a manner that improves- ii. Glucose variability (inter-quartile range)
  IQR is the difference between the 75th and 25th percentiles. Change from baseline was calculated as IQR at baseline minus IQR value at final visit (32 weeks).
Time Frame: baseline to final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
mg/dL | -9 (9.1) | -7.7 (19.4) | -12.1 (14)

6. Secondary Outcome: Change From Baseline in Glucose Exposure (Area Under the Diurnal Median Curve or AUC)
Description: Employ Continuous Glucose Monitoring (CGM) with Ambulatory Glucose Profile (AGP) analysis to characterize the diurnal patterns produced by oral medications (metformin) used in the treatment of type 2 diabetes.
  Employ CGM to measure the effect of exenatide, insulin glargine and exenatide plus insulin glargine in terms of underlying physiological defects and alter medications in a manner that improves- i. Glucose exposure (area under the diurnal median curve) Change from baseline was calculated as area under the diurnal median curve at baseline minus AUC value at final visit (32 weeks).
  AUC is calculated using modified rectangle method AUC = sum of superscript 23, subscript i=0 P subscript 50i I = hour of day P subscript 50i = smoother 50th percentile value for ith hour of day
Time Frame: baseline - final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: mg/dL*24hr
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
mg/dL*24hr | -1207.1 (661.1) | -1476.2 (849.2) | -1315 (953.9)

7. Secondary Outcome: Change From Baseline in Weight Changes
Description: Measure the changes in weight attributable to exenatide, insulin glargine and their combinations.
  Employ CGM with AGP analysis to determine if there is an incremental benefit for subjects who do not reach target to add exenatide to insulin glargine or insulin glargine to exenatide in patients taking metformin.
  Change from baseline was calculated as weight in pounds at baseline minus weight in pounds at final visit (32 weeks).
Time Frame: baseline - final visit (32 weeks)
Measure: Mean (Standard Deviation); unit: lbs (pounds)
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Number analyzed (Participants) | 16 | 17 | 16
lbs (pounds) | -13.5 (10.2) | -0.5 (7.7) | -10.3 (10.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for the 32 weeks subjects actively enrolled in trial
Arm/Group | Exenatide | Insulin Glargine | Exenatide + Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 20/20 | 10/20 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (N=20) | Insulin Glargine (N=20) | Exenatide + Insulin Glargine (N=20)
nausea and vomiting (Gastrointestinal disorders) | 17 (17) | 0 (0) | 0 (0) — 17 subjects on Exenatide experienced nausea and vomiting. All resolved except for 1 subject were it persisted through the end of the study.
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — Allergic reaction
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Itching at the injection sites. Persisted through end of study.
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) — Symptoms resolved on their own.
Hypoglycemia (Endocrine disorders) | 4 (14) | 9 (24) | 13 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No